CLINICAL TRIAL: NCT00687011
Title: Open-label Clinical Trial to Assess the Efficacy, Tolerability and Safety of a Single IV Dose of Palonosetron 0.25 mg + Dexamethasone IV in the Prevention of Moderately Emetogenic Chemotherapy-induced Nausea and Vomit (CINV).
Brief Title: Palonosetron Plus Dexamethasone in Moderately Emetogenic Chemotherapy Induced Nausea and Vomiting (Study P04594)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: P04594
Record Dates: First submitted 2008-05-27; First posted 2008-05-30 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Neoplasms; Nausea; Vomiting
Keywords: Antiemetic
MeSH Terms: conditions — Neoplasms; Nausea; Vomiting | interventions — Palonosetron; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Palonosetron-dexamethasone (Experimental)
  Interventions: Drug: Palonosetron and Dexamethasone

INTERVENTIONS:
Drug: Palonosetron and Dexamethasone — 0.25 mg IV single dose, 30 minutes prior to the administration of the major chemotherapeutic agent, plus single IV dose of dexamethasone 8 mg administered 15 minutes before chemotherapy (in the event of a shortage of IV dexamethasone, a single oral dose of dexamethasone 20 mg or a single IV dose of methylprednisolone 125 mg could be administered).
  Other Names: SCH 734291

SUMMARY:
The purpose of this study is to determine if a single intravenous (IV) dose of palonosetron 0.25 mg plus a single IV dose of dexamethasone 8 mg is effective to prevent nausea and vomiting induced by moderately emetogenic chemotherapy in subjects with cancer.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, >= 18 years of age.
* Histologically or cytologically confirmed malignant disease.
* Naive or non-naive to chemotherapy.
* Karnofsky index >= 70%.
* Scheduled to receive a single dose of at least one of the following agents administered on Study Day 1: any dose of Dactynomicin, Carboplatin, Epirubicin, Idarubicin, Ifosfamide, Irinotecan, Lomustine; or Methotrexate >250 mg/m^2, or Cyclophosphamide <=1500 mg/m^2, or Mitoxantrone <15 mg/m^2, or Doxorubicin >= 20 mg/m^2, or Citarabin > 1g/m^2, Melphalan > 50 mg/m^2 , oxaliplatin > 75 mg/m^2 administered over 1 to 4 hours. The administration of the major chemotherapeutic agent (which is the most emetogenic agent according to the classification of Hesketh, et al., The Oncologist 1999, 4: 191-196) defined Study Day 1 and administration of this agent should not extend beyond 4 hours.
* Provided signed written informed consent.
* Females of childbearing potential must be using reliable contraceptive measures with a negative pregnancy test at the pre-treatment visit.
* If a patient had a known hepatic, renal or cardiovascular impairment and is scheduled to receive the above mentioned chemotherapeutic agents, he/she could be enrolled in this study at the discretion of the investigator.
* If a patient had experienced at maximum mild nausea following any previous chemotherapy regimen, he/she could be enrolled in this study at the discretion of the investigator.

Exclusion Criteria:

* Unable to understand or cooperate with the study procedures.
* Received any investigational drugs within 30 days before study entry.
* Received any drug with potential anti-emetic efficacy within 24 hours of the start of treatment or will be scheduled to receive until Study Day 5 including 5-HT3 receptor antagonists, metoclopramide, phenothiazine anti-emetics (including prochlorperazine, thiethylperazine and perphenazine), scopolamine, diphenhydramine, chlorpheniramine maleate, trimethobenzamide, all benzodiazepines except temazepam or triazolam used once nightly for sleep, haloperidol, droperidol, tetrahydrocannabinol, or nabilone, any corticosteroid including dexamethasone, hydrocortisone, methylprednisolone, prednisone (excluding topical or inhaled preparations).
* Seizure disorder requiring anticonvulsant medication unless clinically stable and free of seizure activity.
* Experienced any vomiting, retching, or NCI Common Toxicity Criteria grade 2 or 3 nausea in the 24 hours preceding chemotherapy.
* Ongoing vomiting from any organic etiology.
* Experienced nausea (moderate or severe) or vomiting following any previous chemotherapy. At the discretion of the investigator, a patient who experienced at maximum mild nausea following any previous chemotherapy might not be excluded from this study.
* Scheduled to receive any dose of cisplatin, carmustine, hexametilamine, dacarbazine, Mecloretamine, Streptozotocin, Procarbazine o Cyclophosphamide > 1500 mg/m^2 or any other chemotherapeutic agent with an emetogenicity level 5 according to the classification of NCCN Guidelines v1 2005 during Study Days 2-6.
* Known contraindication to 5-HT3 receptor antagonists.
* Scheduled to receive radiotherapy of the upper abdomen or cranium during Study Day 2-6.
* QTc > 500 msec at baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2006-10-10 (Actual); Primary Completion 2008-10-27 (Actual); Study Completion 2008-10-27 (Actual)

PRIMARY OUTCOMES:
Proportion of patients having achieved complete response (CR), defined as no emetic episodes and no rescue medication. | During 24 hours after administration of chemotherapy.

SECONDARY OUTCOMES:
Proportion of patients who achieved a CR and of those who achieved complete control; Number of emetic episodes; Time to first emetic episode, to administration and need for rescue therapy; and to treatment failure | Days 1 to 5 at different time intervals for each secondary outcome.
Severity of nausea; Patient global satisfaction; Quality of life questionnaire | Days 1 to 5 at different time intervals for each secondary outcome.

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html